CLINICAL TRIAL: NCT04438044
Title: A Phase II, Multicenter, Open-label Study to Evaluate the Safety and Efficacy of ICP-022 in Patients With Recurrent/Refractory Central Nervous System Lymphoma and Recurrent/Refractory Secondary Central Nervous System Lymphoma
Brief Title: A Study to Evaluate ICP-022 in Patients With R/R PCNSL and SCNSL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00106
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: PCNSL; Secondary Central Nervous System Lymphoma
Keywords: Recurrent or refractory
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICP-022 (Experimental): 150mg,QD
  Interventions: Drug: ICP-022

INTERVENTIONS:
Drug: ICP-022 — ICP-022 The drug product is a white, round, uncoated tablet

SUMMARY:
The phase II clinical study is to investigate the safety, tolerability, efficacy and pharmacokinetics of ICP-022.

DETAILED DESCRIPTION:
Safety, tolerability evaluation, and anti-tumor effects of ICP-022 in Chinese patients with Recurrent/Refractory Central Nervous System Lymphoma (PCNSL) and Recurrent/Refractory Secondary Central Nervous System Lymphoma (SCNSL) will be evaluated in approximately 82 subjects. Pharmacokinetics of ICP-022 will be evaluated in approximately 20 subjects .

ELIGIBILITY:
Key Inclusion Criteria:

1. Men and women ≥ 18, and ≤75 years of age
2. Histologically documented PCNSL, or histologically documented systemic diffuse large B-cell lymphoma (DLBCL) for SCNSL.
3. Subjects with refractory or relapsed disease, one prior CNS directed therapy, and ≤ 4 systemic treatments.
4. ECOG performance status of 0-2
5. Able to provide signed written informed consent

Key Exclusion Criteria:

1. Patients with SCNSL actively receiving treatment for extra-CNS disease are excluded
2. T-cell lymphoma.
3. Patient requires more than 8 mg of dexamethasone daily or the equivalent.
4. Non-hematological toxicity must recover to ≤ Grade 1 from prior anti-cancer therapy (except for alopecia)
5. Known active infection with HBV, HCV or HIV.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The efficacy measured by overall response rate (ORR) | Cycle 1-6 once every 2 cycles; more than 6 cycles once every 3 cycles. Each cycle is 28 days

SECONDARY OUTCOMES:
The occurrence of adverse events and serious adverse events | every cycle, first cycle every week. Each cycle is 28 days
  The safety of ICP-022 measured by the occurrence of adverse events and serious adverse events according to NCI-CTCAE 4.03 grading criteria
The efficacy measured by progression free survival (PFS) | cycle 1-6 once every 2 cycles; more than 6 cycles once every 3 cycles. Each cycle is 28 days
The efficacy measured by duration of response (DOR) | cycle 1-6 once every 2 cycles; monre than 6 cycles once every 3 cycles. Each cycle is 28 days

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Capital Medical University Xuanwu Hospital, Beijing, Beijing Municipality
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No